# Skin Care Trials - Evaluating Patient Experiences in Skin Care Clinical Studies

A Participant Agreement Form for Power Clinical Trial's
Observational Clinical Trial: Understanding Your Rights and
Responsibilities

Date: February 10, 2023

Important Details About the Informed Consent Form

You have been identified as a potential participant in a clinical study observing patients following skin care routines. This form provides comprehensive information about the study, including its purpose, methodology, potential benefits, and risks.

Before making a decision to participate, it is recommended that you seek advice from trusted individuals and take the necessary time to consider your options. If there is anything unclear in this document, please do not hesitate to speak with the researcher for clarification.

The Purpose of This Skin Care Clinical Trial

Skin care refers to the various practices and products used to maintain the health and appearance of the skin. This includes cleansing, moisturizing, protecting from sun damage, and treating skin conditions such as acne, wrinkles, and dark spots.

Skin care clinical trials are conducted to evaluate the safety and efficacy of new skin care products and treatments. They play an important role in advancing our understanding of skin care and the development of new and improved products.

By participating in a clinical trial, individuals can help to contribute to the advancement of skin care and improve the quality of life for people with skin concerns.

The objective of this clinical study is to observe patients who are undergoing skin care routines and analyze their patterns of completion and withdrawal rates during participation in an unrelated medical intervention clinical trial.

### Observational Clinical Trial: A Deeper Look

In this medical trial, you will be participating in an observational study, which is a type of clinical trial that involves observing individuals without recommending any specific treatments or interventions.

The primary goal of this study is to gather information about the outcomes of individuals who are diagnosed with a particular condition, without making any changes to their current care plan. By participating in this study, you will be helping researchers gain valuable insights into the natural progression of the condition and better understand its effects on the individuals who have it.

## Skin Care Trials Comparison

It's important to note that there are many other types of clinical trials for skin care that are interventional in nature, meaning that you would have to undergo a specific treatment if you participate in those studies.

To help you make an informed decision, you can research and compare different clinical trials by reading medical journals and other trusted sources of information. A good place to start is clinicaltrials.gov, which lists a wide range of <u>skin care studies</u>, as well as Power's website, which has information about various <u>skin care clinical trials</u>.

# Gathering Information About Clinical Trial Experiences

As a participant in this clinical trial, you will be asked to share information about your experiences. To gather this information, you will be asked to complete a questionnaire every two weeks.

The questionnaire is relatively straightforward and should take approximately 20-30 minutes to complete. Additionally, you will have check-in calls with the study team on a quarterly basis for as long as you continue to participate in the trial.

It's important to note that your participation in this aspect of the trial is entirely voluntary. You are free to decline to answer any or all questions, and you can choose to discontinue your involvement in the trial at any time. Your participation in this trial is important to us, and we are committed to ensuring that you feel comfortable and respected throughout the process.

Your anonymity will be maintained throughout the entire clinical trial experience. To ensure this, please do not include any personal or identifying information in your responses to the questionnaires.

The research team will take all necessary measures to protect your confidentiality. However, it should be noted that there may be certain legal circumstances in which the researcher is obligated to disclose your information.

#### Risks

The importance of patient safety and well-being is a top priority in any clinical trial.

However, when it comes to interventional trials where participants are receiving new treatments, there is a risk that unintended side effects may occur. In our observational clinical trial, participants are not receiving any new treatments, and therefore, the risk of negative health outcomes is greatly reduced, if not entirely eliminated.

Protecting the privacy of participant information is a critical aspect of any clinical trial. In our medical study, every effort has been made to minimize the risk of a breach of confidentiality. All data collected from participants are anonymous, and access to this information is restricted to the research team only.

The storage of all records, including call logs, online transactions, forms, and surveys, has been secured with the use of encryption and password protection to ensure the privacy of participant information.

#### Benefits

While participating in this clinical trial may not offer direct benefits to individuals, your contribution can significantly shape the future of skin care treatments.

The data gathered from the participants will help researchers better understand enrolment patterns, identify possible challenges, and provide insights that can improve the enrolment process for future skin care patients. As such, your participation in this clinical trial will be a valuable contribution to the advancement of medical research.

# Read More on Representation in Clinical Trials

Finding information on representation in clinical trials can be difficult, but there are several online resources available that can help. To assist you in your research, here are some suggested sources you may want to consider exploring:

Westen, Drew I., Shannon Wiltsey Stirman, and Robert J. DeRubeis. "Are research patients and clinical trials representative of clinical practice?." (2006).

Tao, Cui, Guoqian Jiang, Weiqi Wei, Harold R. Solbrig, and Christopher G. Chute.
"Towards semantic-web based representation and harmonization of standard meta-data models for clinical studies." *AMIA summits on translational science proceedings* 2011 (2011): 59.

#### Consent

I have meticulously perused this document, either by myself or with the assistance of someone else who has read it to me.

I have a complete understanding of the information contained within and have been given the chance to pose any inquiries I may have had. I acknowledge that my participation in this study is purely optional and that I am at liberty to terminate my involvement at any moment without having to give an explanation and without incurring any fees. I am aware that I will be given a duplicate of this informed consent form.

| I wholeheartedly consent to taking part in | this research project. |
|---|---|
| Printed Name of Participant | |
| Participant Signature | |
| Date | |
| Declaration of Person Taking Conse | ent |
| During the review process of this skin care participant was fully informed of its purpos | e clinical trial document, I ensured that the se, procedures, and potential outcomes. |
| a complete understanding of the informati | ey may have had and made sure that they had on presented. It is important to stress that the irely optional and they can choose to withdraw uences or fees. |
| The participant has given their informed control provided to them for their records after the | • • |
| Drinted Name of Derson Taking Conser | |
| Printed Name of Person Taking Consei | ıt |
| Signature of Person Taking Consent | |
| Date | |